CLINICAL TRIAL: NCT03399318
Title: Aggressive Antipyretics in CNS Malaria: A Randomized-Controlled Trial Assessing Antipyretic Efficacy and Parasite Clearance Effects
Brief Title: Aggressive Antipyretics for Fever Reduction in CNS Malaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Gretchen Birbeck, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RSRB00067717; R01NS102176 (NIH)
Record Dates: First submitted 2017-10-17; First posted 2018-01-16 (Actual); Results first posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Malaria; Seizures; Coma; Parasitemia; Hyperpyrexia; Fever
Keywords: HRP2
MeSH Terms: conditions — Malaria; Seizures; Coma; Parasitemia; Hyperthermia; Fever | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aggressive Antipyretics (Experimental): regardless of temperature, children allocated to this arm will receive acetaminophen (30 milligrams (mg)/ kilogram (kg) load then 15mg/kg Q6 hours) and ibuprofen (10mg/kg Q 6 hours) for 72 hours. Pediatric syrup formulations of both agents will be administered orally or via nasogastric tube. For temperatures over 38.5 degrees Celsius, placebo will be added and if the fever persists, a cooling fan will be added.
  Interventions: Drug: Acetaminophen; Drug: Ibuprofen
- Usual Care (Placebo Comparator): will receive placebo for acetaminophen and placebo for ibuprofen. If they have a temperature over 38.5 degrees Celsius, they will receive acetaminophen (15mg/kg, Q6 hours), as needed. If the fever persists, a cooling fan will be added.
  Interventions: Drug: placebo for acetaminophen; Drug: placebo for ibuprofen

INTERVENTIONS:
Drug: Acetaminophen — 30 mg/kg load then 15mg/kg Q6 hours for the Aggressive Antipyretic Arm
  Acetaminophen is also given to children in the placebo arm when they have a fever over 38.5 degrees Celsius during scheduled clinical assessments
  Other Names: Paracetamol
  Arms: Aggressive Antipyretics
Drug: Ibuprofen — 10 mg/kg Q6 hours for the Aggressive Antipyretic Arm
  Other Names: Brufen
  Arms: Aggressive Antipyretics
Drug: placebo for acetaminophen — placebo for acetaminophen for children in the Usual Care arm
  For children in the Aggressive Antipyretic Arm, when they have a temperature over 38.5 degrees Celsius they are treated with a placebo
  Other Names: Placebo
  Arms: Usual Care
Drug: placebo for ibuprofen — placebo for ibuprofen
  Other Names: Placebo
  Arms: Usual Care

SUMMARY:
The study will examine whether prophylactic and scheduled treatment with acetaminophen and ibuprofen can decrease the maximum temperature experienced during the acute illness in children with CNS malaria.

DETAILED DESCRIPTION:
Despite ongoing eradication efforts, malaria remains a major public health challenge in Africa where annually, ~250,000 children with malaria experience a neurologic injury with subsequent neurodisability. In other central nervous system (CNS) disorders, fever is a recognized cause of worsening secondary neurologic injury and ex-tensive efforts are made to avoid hyperthermia or induce hypothermia for neuroprotection. Evidence indicates that among children with CNS malaria a higher temperature during the acute illness is a risk factor for post-infectious neurologic sequelae. As such, aggressive antipyretic therapy may be warranted, at least among children with complicated malaria who are at substantial risk of brain injury. Previous clinical trials conducted primarily in children with uncomplicated malaria and using only a single antipyretic medication have shown limited benefits in terms of fever reduction; however, no studies to date have examined malaria fever management using dual therapies. Enthusiasm for aggressive fever reduction measures among clinicians caring for children with malaria has been curbed by in vitro findings that malaria parasite replication slows at higher temperatures and a single clinical trial in which peripheral parasite clearance was slower in children receiving treatment for fever. However, the relationship between temperature and malaria parasite behavior is complex. Additional in vitro data suggest that at febrile temperatures uninfected red blood cells (RBCs) are more likely to adhere to infected RBCs, worsening the process of sequestration, increasing the parasite burden obstructing microvascular cerebral blood flow, and perhaps contributing to ongoing immunopathogenesis in CNS malaria. In this exploratory clinical trial of aggressive antipyretic therapy, children hospitalized with CNS malaria will be randomized to usual care (acetaminophen every 6 hours for a temperature ≥ 38.5ºC) vs. prophylactic acetaminophen and ibuprofen every 6 hours for 72 hours. This proof-of-concept study will determine whether aggressive antipyretic therapy results in a lower mean maximum temperature relative to usual care. Serial quantitative levels of histidine rich protein 2 (HRP2), a P. falciparum-specific protein that facilitates estimates of whole body parasite burden and CNS parasite sequestration, will also be collected to clarify the relationship between antipyretic use and in vivo parasite behavior. Findings from this study will determine whether a Phase III clinical trial of aggressive antipyretics for neuroprotection in pediatric CNS malaria should be undertaken. This study will take place in Zambia and Malawi, where prior NIH-funded collaborations have assisted in developing the substantial infrastructure needed to undertake a clinical trial of this nature.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of Plasmodium falciparum malaria infection by peripheral blood smear or rapid diagnostic test
* Central nervous system (CNS) symptoms associated with malaria. CEREBRAL MALARIA (CM): Impaired consciousness with a Blantyre Coma Score (BCS)(73) ≤2 in children under 5 years or a Glasgow Coma score (GCS) ≤10 in children ≥5 years OR CNS MALARIA: Complicated seizure(s), meaning prolonged (>15 minutes), focal or multiple; or impaired consciousness or other evidence of impaired consciousness (confusion, delirium) without frank coma (BCS>2, GCS =11-14)

Exclusion Criteria:

* Circulatory failure (cold extremities, capillary refill > 3 seconds, sunken eyes, ↓ skin turgor)
* Vomiting in the past 2 hours
* Serum creatinine (Cr) > 1.2 mg/dL
* A history of liver disease
* Jaundice or a total bilirubin of >3.0mg/dL
* A history of gastric ulcers or gastrointestinal bleeding
* A history of thrombocytopenia or other primary hematologic disorder
* Petechiae or other clinical indications of bleeding abnormalities
* A known allergy to ibuprofen, acetaminophen, aspirin or any non-steroidal medication
* Any contraindication for nasogastric tube (NGT) placement and/or delivery of enteral medications

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 256 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen L Birbeck, MD, Principal Investigator — University of Rochester
Locations (3):
- Pediatric Research Ward at Queen Elizabeth Central Hospital, Blantyre, Malawi
- Zambia (2):
  - Chipata Central Hospital, Chipata, Eastern Province
  - University Teaching Hospital's Lusaka Childrens Hospital, Lusaka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Birbeck GL, Seydel KB, Mwanza S, Tembo D, Chilombe M, Watts A, Ume-Ezeoke I, Mathews M, Patel AA, Mwenechanya M, Pensulo P, McDermott MP. Acetaminophen and Ibuprofen in Pediatric Central Nervous System Malaria: A Randomized Clinical Trial. JAMA Neurol. 2024 Aug 1;81(8):857-865. doi: 10.1001/jamaneurol.2024.1677. PMID 38857015
- [Derived] Tembo D, Mwanza S, Mwaba C, Dallah I, Wa Somwe S, Seydel KB, Birbeck GL. Risk factors for acute kidney injury at presentation among children with CNS malaria: a case control study. Malar J. 2022 Nov 1;21(1):310. doi: 10.1186/s12936-022-04327-y. PMID 36316704

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in Malawi and Zambia from 2019 to 2022. In Malawi, enrolment occurred at Queen Elizabeth Central Hospital in Blantyre. In Zambia, the trial was conducted at the University Teaching Hospital in Lusaka and Chipata Central Hospital in the Eastern Province. This work was approved by the appropriate ethics review boards in Zambia and Malawi and at the University of Rochester in the United States.
Groups:
- Aggressive Antipyretics (AA): AA children received a loading dose of acetaminophen (30 mg/kg) followed by 15 mg/kg every 6 hours regardless of clinical temperature for 72 hours. No loading dose was given if an antipyretic had been administered in the past 24 hours. In addition, AA children received ibuprofen 10mg/kg Q6 hours for 72 hours. A cooling fan was added for anyone with persistent fevers. When T≥38.5°C was detected, 15 mg/kg of placebo was added in the AA group.
- Usual Care (UC).: UC children received 15 mg/kg of acetaminophen as needed every 6 hours for T≥38.5°C based upon clinical axillary temperatures obtained every 2 hours in Malawi and every 6 hours in Zambia. No loading dose was given if an antipyretic had been administered in the past 24 hours. To maintain double-blinding, an initial loading dose of placebo and placebos for acetaminophen and ibuprofen were used in the UC group.
Period: Overall Study
Arm/Group | Aggressive Antipyretics (AA) | Usual Care (UC).
Started | 128 | 128
Completed | 128 | 128
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible children were 24-132 months of age with evidence of P. falciparum infection, based upon a thick peripheral blood smear or rapid diagnostic test, and symptoms of CNS malaria including complicated seizures (multiple seizures, focal seizures or prolonged seizures lasting more than 15 minutes) or impaired consciousness
Groups:
- Total: Total of all reporting groups
Arm/Group | Aggressive Antipyretics (AA) | Usual Care (UC). | Total
Number analyzed (Participants) | 128 | 128 | 256
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 4.4 [2.9 to 6.6] | 3.8 [2.8 to 5.1] | 4.1 [2.9 to 5.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 56 | 115
  Male | 69 | 72 | 141
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 128 | 128 | 256
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Malawi | 74 | 72 | 146
  Zambia | 54 | 56 | 110
Weight [Mean (Standard Deviation); unit: units on a scale - kg] | 15.1 (4.4) | 14.0 (3.2) | 14.6 (3.8)
Admission temperature [Mean (Standard Deviation); unit: degrees of Celsius (°C)] | 38.1 (1.3) | 38.1 (1.3) | 38.1 (1.3)
Cerebral malaria [Count of Participants; unit: Participants] | 83 | 72 | 155
Blantyre Coma Score [Count of Participants; unit: Participants] — BSC is ordinal 0-5 with 0 being worst and 5 being best (i.e. normal)
  Participants
    0 | 2 | 6 | 8
    1 | 22 | 27 | 49
    2 | 48 | 50 | 98
    3 | 21 | 16 | 37
    4 | 12 | 11 | 23
    5 | 23 | 18 | 41
Seizures [Number; unit: participants] — Seizures were captured by bedside convulsion charts and a 30-minute EEG obtained daily until return to consciousness. Seizures were categorized as none, single and brief, or multiple or prolonged, yielding a three-category outcome. Population: One research file was lost and these data were not otherwise recoverable.
  participants
    None: number analyzed (Participants) | 127 | 128 | 255
    None | 23 | 20 | 43
    Single and brief: number analyzed (Participants) | 127 | 128 | 255
    Single and brief | 16 | 10 | 26
    Multiple or prolonged: number analyzed (Participants) | 127 | 128 | 255
    Multiple or prolonged | 88 | 98 | 186
Had received antipyretics [Number; unit: participants] | 115 | 110 | 225
Had received anticonvulsant [Count of Participants; unit: Participants] | 64 | 69 | 133
Quantative parasite count [Geometric Mean (Inter-Quartile Range); unit: parasite per microliter] — Population: Quantitative counts are only applicable to participants who had parasite in their blood. Those who were smear negative on enrolment due to rapid antimalairal administration were not included in the analysis. These individuals had their diagnosis confirmed by a rapid diagnostic test
  parasite per microliter
    number analyzed (Participants) | 92 | 89 | 181
    (all) | 3281 [280 to 93075] | 1890 [160 to 45000] | 2100 [210 to 84500]
HRP2-(ng/ml) [Geometric Mean (Inter-Quartile Range); unit: ng/ml] | 123 [9 to 424] | 86 [5 to 376] | 108 [8 to 400]
Packed Cell Volume [Mean (Standard Deviation); unit: percent - %] — The packed cell volume (PCV) is a measurement of the proportion of blood that is made up of cells
  percent - % | 28 (7) | 29 (7) | 29 (7)
Creatinine [Mean (Standard Deviation); unit: units on a scale - mg/dL] | 0.64 (0.23) | 0.63 (0.20) | 0.64 (0.22)
HIV Positive [Count of Participants; unit: Participants] | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Mean Maximum Temperature
Description: Mean maximum temperature (Tmax). Tmax will be defined as the highest temperature during the study duration (72 hours) in degrees Celsius recorded by a continuous temperature monitor.
  The continuous temperature monitors are not magnetic resonance imaging (MRI) compatible. If TMAX is a clinical temperature obtained when continuous monitoring data is not available, the clinical TMAX will be used as the primary outcome.
Time Frame: 72 hours
Measure: Mean (95% Confidence Interval); unit: degrees of Celsius
Arm/Group | Aggressive Antipyretics (AA) | Usual Care (UC).
Number analyzed (Participants) | 128 | 128
degrees of Celsius | 38.6 [38.4 to 38.7] | 39.2 [39.1 to 39.3]
Statistical Analysis 1: Comparison: Aggressive Antipyretics (AA) vs Usual Care (UC); The analysis of the primary outcome variable, Tmax, involved fitting an analysis of 206 covariance model with treatment group as the factor of interest, country and disease severity 207 (CM=yes, no) as stratification factors, and admission temperature as a covariate. The estimated 208 treatment effect and associated 95% confidence interval, as well as a t-test for significance of the treatment effect, were derived from this model; Test type: Superiority; p < 0.0001, t-test, 2 sided — treatment group as the factor of interest, country and disease severity 207 (CM=yes, no) as stratification factors, and admission temperature as a covariate. A t-test for significance of the treatment effect, were derived from this model

2. Primary Outcome: Seizure Severity
Description: Seizures were categorized as none, single and brief, or multiple or prolonged, yielding a three-category outcome.
Time Frame: 72 hours
Population: One research file was lost and these data were not otherwise recoverable
Measure: Count of Participants; unit: Participants
Arm/Group | Aggressive Antipyretics (AA) | Usual Care (UC).
Number analyzed (Participants) | 127 | 128
Participants
  None | 107 | 88
  Single and brief | 10 | 6
  Multiple or Prolonged | 10 | 34
Statistical Analysis 1: Comparison: Aggressive Antipyretics (AA) vs Usual Care (UC); Seizure occurrence defined as a three-level ordinal variable was analyzed using a 223 multinomial logistic regression model because there was evidence that the proportional odds 224 assumption did not hold. This model included treatment group as the factor of interest and 225 country and disease severity as stratification factors. The adjusted treatment group odds ratio, 226 and its associated 95% confidence interval were derived from this model; Test type: Superiority; p < 0.05, Regression, Logistic; Odds Ratio (OR) = 0.09, 95% CI 2-sided [.03 to .27]

3. Secondary Outcome: Parasite Clearance
Description: Parasite clearance was based upon AUC for plasma HRP2 concentration every six hours
Time Frame: 72 hours
Population: Exclusion of 38 children with missing data
Measure: Median (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Aggressive Antipyretics (AA) | Usual Care (UC).
Number analyzed (Participants) | 108 | 110
ng*hr/mL | 86.3 [78.2 to 94.4] | 80 [71.5 to 88.4]
Statistical Analysis 1: Comparison: Aggressive Antipyretics (AA) vs Usual Care (UC); Parasite clearance measured by log10 (HRP2 level) was analyzed with a repeated 228 measures analysis of covariance model (mixed model repeated measures)35 with terms for 229 treatment group, country, disease severity, log10(HRP2 level) at admission, time (treated as a 230 categorical variable), and interaction terms for admission log10(HRP2 level) and time, and for 231 treatment group and time; Test type: Superiority; p < 0.05, ANCOVA — The covariance matrix for the within-participant observations was 232 modeled using an unstructured pattern; Time to parasite clearance was 235 evaluated using a discrete-time proportional hazards model with a complementary log-log link; Odds Ratio, log = 6.3, 95% CI 2-sided [-5.1 to 17.7] — The adjusted treatment group difference in mean area 233 under the log10(HRP2 level) × time curve was estimated using appropriate contrasts among the 234 treatment group means over time that quantify this comparison; The model included terms for treatment group, country, and disease severity

4. Secondary Outcome: Area-under-the-curve (AUC) of Fever ≥ 38.5°C (Best)
Description: AUC fever for temperatures above 37.5 degrees Celsius based upon continuous temperature monitoring A secondary efficacy measure included fever exposure as measured by the area under the temperature × time curve for T≥38.5°C during the 72-hour follow-up period, categorized as 0, > 0 and < 2, and ≥ 2 degree-hours. An ordinal logistic regression model assuming proportional odds with terms for treatment group, country, and disease severity as covariates was used to derive the estimated adjusted treatment group odds ratio and associated 95% confidence interval. Sensitivity analyses with best-case and worst-case imputation were performed to accommodate missing data for the 12 participants with insufficient temperature data to determine the proper outcome category
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Aggressive Antipyretics (AA) | Usual Care (UC).
Number analyzed (Participants) | 128 | 128
Participants
  0 | 67 | 37
  > 0 and < 2 | 47 | 54
  ≥ 2 | 14 | 37
Statistical Analysis 1: Comparison: Aggressive Antipyretics (AA) vs Usual Care (UC); A secondary efficacy measure included fever exposure as measured by the area under 214 the temperature × time curve for T≥38.5°C during the 72-hour follow-up period, categorized as 215 0, > 0 and < 2, and ≥ 2 degree-hours; Test type: Superiority; p < 0.05, Regression, Logistic — An ordinal logistic regression model assuming 216 proportional odds with terms for treatment group, country, and disease severity as covariates was used to derive the estimated adjusted treatment group odds ratio and 95%CI; Sensitivity analyses with best-case and worst-case imputation were 219 performed to accommodate missing data; Odds Ratio (OR) = .32, 95% CI 2-sided [.20 to .52]

ADVERSE EVENTS:
Time Frame: 72 hours
Arm/Group | Aggressive Antipyretics (AA) | Usual Care (UC).
All-Cause Mortality (participants affected / at risk) | 3/128 | 10/128
Serious Adverse Events (participants affected / at risk) | 15/128 | 25/128
Other Adverse Events (participants affected / at risk) | 102/128 | 87/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aggressive Antipyretics (AA) (N=128) | Usual Care (UC). (N=128)
Death (General disorders) | 3 (3) | 10 (10)
Any bleeding (Vascular disorders) | 0 (0) | 1 (1)
Clinical signs of bleeding (Vascular disorders) | 0 (0) | 1 (1)
Creatinine increase (Renal and urinary disorders) | 3 (5) | 0 (0)
Neurologic deficits at discharge (Nervous system disorders) | 9 (9) | 10 (10)
Shock (General disorders) | 0 (0) | 1 (1)
Shock with necrotic digits (Vascular disorders) | 0 (0) | 1 (1)
Status epilepticus and prolonged apnea (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aggressive Antipyretics (AA) (N=128) | Usual Care (UC). (N=128)
Any bleeding (Vascular disorders) | 17 (18) | 9 (10)
Clinical signs of bleeding (Vascular disorders) | 5 (5) | 2 (2)
Creatinine increase (Renal and urinary disorders) | 61 (100) | 48 (81)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Elevated lactate (Metabolism and nutrition disorders) | 12 (18) | 19 (24)
Fell from bed (General disorders) | 2 (2) | 2 (2)
Hyperbilirubinemia (Hepatobiliary disorders) | 64 (144) | 66 (150)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Misc. lab change (General disorders) | 0 (0) | 1 (1)
Nasogastric tube injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bleeding occult (Blood and lymphatic system disorders) | 12 (13) | 7 (8)
Drop in level of consciousness (General disorders) | 1 (1) | 0 (0) — Participant level of consciousness dropped from BCS 5/5 to BCS 4/5.
Prolonged hospitalization. (Nervous system disorders) | 0 (0) | 1 (1)
Systemic allergic reaction (General disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vomiting (General disorders) | 10 (12) | 9 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT03399318/Prot_SAP_003.pdf
  • Informed Consent Form: Zambian Consent Form (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/18/NCT03399318/ICF_004.pdf
  • Informed Consent Form: Malawian Consent Form (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/18/NCT03399318/ICF_005.pdf